CLINICAL TRIAL: NCT03882489
Title: Estimation of Effective Dose 95 (ED95) of Intrathecal Isobaric 2-chloroprocaine (2-CP) Based on the Height (cm) of a Patient Undergoing Ambulatory Knee Arthroscopy : Dose-finding Study Based on the Continual Reassessment Method (CRM)
Brief Title: Estimation of Effective Dose 95 (ED95) of Intrathecal Isobaric 2-chloroprocaine (2-CP) Based on the Height (cm) of a Patient Undergoing Ambulatory Knee Arthroscopy
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Collaborators: Hôpital de Braine-l'Alleud (Other)
Responsible Party: Sponsor
Other Study IDs: B076201836762
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Knee Arthroscopy
Keywords: spinal anesthesia; Knee Arthroscopy; Chloroprocaine; Height; Effective Dose (ED95); Continual Reassessment Method (CRM)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1 : Height 150-165 cm: Dose-finding study with 4 subjects per dose and a maximum of 40 patients by cohort. The cohort 1 includes patients whose the height is between 150 and 165 cm. To identify the dose to give for reaching the ED95 (effective dose for 95% subjects), isobaric 2-chloroprocaine will be administrated at the dose initial of 40 mg in the cohort 1 for the first 4 subjects. For the next subjects, the doses to administrate will vary 5 mg (0.5 ml) and will be determined by the Continual Reassessment Method (CRM) according to the observed responses in the previous subjects. Doses will be staggered from 25 to 50 mg for cohort 1.
  Interventions: Drug: Isobaric 2-chloroprocaine
- Cohort 2 : Height 166-180 cm: Dose-finding study with 4 subjects per dose and a maximum of 40 patients by cohort. The cohort 2 includes patients whose the height is between 166 and 180 cm. To identify the dose to give for reaching the ED95 (effective dose for 95% subjects), isobaric 2-chloroprocaine will be administrated at the dose initial of 45 mg in the cohort 2 for the first 4 subjects. For the next subjects, the doses to administrate will vary 5 mg (0.5 ml) and will be determined by the Continual Reassessment Method (CRM) according to the observed responses in the previous subjects. Doses will be staggered from 30 to 55 mg for cohort 2.
  Interventions: Drug: Isobaric 2-chloroprocaine
- Cohort 3 : Height 181-195 cm: Dose-finding study with 4 subjects per dose and a maximum of 40 patients by cohort. The cohort 3 includes patients whose the height is between 166 and 180 cm. To identify the dose to give for reaching the ED95 (effective dose for 95% subjects), isobaric 2-chloroprocaine will be administrated at the dose initial of 50 mg in the cohort 3 for the first 4 subjects. For the next subjects, the doses to administrate will vary 5 mg (0.5 ml) and will be determined by the Continual Reassessment Method (CRM) according to the observed responses in the previous subjects. Doses will be staggered from 35 to 60 mg for cohort 3.
  Interventions: Drug: Isobaric 2-chloroprocaine

INTERVENTIONS:
Drug: Isobaric 2-chloroprocaine — The doses of isobaric 2-chloroprocaine will be administrated intrathecally and will be adjusted according to the observed responses in the previous subjects.
  Other Names: Ampres 10mg/ml

SUMMARY:
In ambulatory surgery, the choice of the local anesthetic used is essential. The ideal local anesthetic must allow a quick installation of the spinal block, a duration of the sensory block adapted to the surgery with a minimum of side effects. These side effects include bradycardia, hypotension and block failure during the intraoperative period; bladder retention, transient neurological disorders during the post-operative period. The achievement of kinetic objectives associated with a reduction in side effects is related to the choice of local anesthetic and the dose administered. However, there are interindividual pharmacokinetic variations that make it difficult to predict the effective dose and the unfortunate occurrence of side effects.

In this context, the height of the patient is a criterion involved in the level, the duration of the sensitive motor block and therefore the side effects

The local anesthetic of the amino ester family, isobaric 2-chloroprocaine (2-CP) has been successfully used for spinal anesthesia since several decades. With a short duration of action, it is preferred to other anesthetics for the short-term outpatient surgeries. However, the effective dose 95 (ED95) of intrathecal isobaric 2-CP is currently unknown.

The purpose of this prospective study is to determine the ED95 of the spinal 2-CP using the continuous re-evaluation method (Continual Reassessment Method) (CRM) based on patient's height

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* scheduled outpatient knee arthroscopy
* between 18 and 80 years old
* American Society of Anesthesiologists physical status (ASA) < III
* Height between 150 and 195 cm

Exclusion Criteria:

* cardiac pathology (such as heart failure, aortic stenosis)
* coagulation disorder (International Normalized Ratio (INR) > 1.3, platelets<80.000/mm3)
* known allergy to local anaesthetics
* central and peripheral neuropathies
* patient's refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing ambulatory knee arthroscopy under the spinal anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-17 (Actual)

PRIMARY OUTCOMES:
Success or failure of anesthesia | perioperative
  The anesthesia will be considered as a success if there is an extension of the sensory block to the Th12 dermatome after inflation of the tourniquet, absence of pain during tourniquet inflation, incision and overall surgery.
  Or the anesthesia will be considered as a failure if there is an absence of extension of the sensory block at the Th12 dermatome, pain at the tourniquet inflation, at the incision, or during surgery.

SECONDARY OUTCOMES:
Maximum level of sensory block assessed as loss of sensation to pinprick, cold | Until complete release of sensory block (up to 5 hours after surgery)
  The level of sensory block will be assessed as loss of sensation to pinprick and cold at 5, 10, 20 and 30 minutes after the intrathecal injection (corresponding to time 0), every 10 minutes in the Post Anesthesia Care Unit (PACU) and every 30 minutes after PACU discharge.
Level of motor block assessed by the Bromage score | Until complete release of motor block (up to 5 hours after surgery)
  The level of motor block will be determined at 5, 10, 20 and 30 minutes after intrathecal injection (corresponding to time 0) and every 10 minutes in the post-anesthesia care unit (PACU). The level of motor block will be assessed by using the Bromage Scale.
Side-effects (nausea, vomiting) | up to 5 hours after surgery
  Nausea and vomiting are treated in the PACU and the post operative unit.
Pain as assessed by Visual Analog Scale | up to 24 hours after surgery
  Pain levels will be determined at tourniquet inflation, incision, every 10 minutes in the post-anesthesia care unit (PACU), every 30 minutes after PACU discharge and 24h after the surgery at home (by phone). Visual Analog pain score (scale = 0 no pain; 10= worst pain imaginable)
End time of sensory block | Until complete release of sensory block (up to 5 hours after surgery)
  The patient is asked to note the time at which he/she feels that he/she has regained a strictly normal sensitivity
Time to void | up to maximum 5 hours after surgery
  The time to obtain the first micturition will be noted.
Bladder volume before first micturition | up to maximum 5 hours after surgery
  An evacuating bladder catheterization is performed when a bladder volume greater than 600 mL, confirmed by a Bladderscan device, is associated with the following signs and/or symptoms: hypogastric pain, anuria or overflow urination.
Time to eligibility for discharge defined by complete regression of sensory block | up to maximum 5 hours after surgery
  Time of discharge of the patient from the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Guntz, MD, PhD, Principal Investigator — Université Libre de Bruxelles (ULB), Braine-l'Alleud Hospital; Emmanuel Guntz, Principal Investigator — Université Libre de Bruxelles (ULB), Braine-l'Alleud Hospital
Locations (1):
- Braine-l'Alleud Hospital, Braine-l'Alleud, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yu X, Zhang F. The effect of parturient height on the median effective dose of intrathecally administered ropivacaine. Ann Saudi Med. 2016 Sep-Oct;36(5):328-333. doi: 10.5144/0256-4947.2016.328. PMID 27710984
- [Background] Forster JG, Rosenberg PH, Harilainen A, Sandelin J, Pitkanen MT. Chloroprocaine 40 mg produces shorter spinal block than articaine 40 mg in day-case knee arthroscopy patients. Acta Anaesthesiol Scand. 2013 Aug;57(7):911-9. doi: 10.1111/aas.12107. Epub 2013 Mar 25. PMID 23521140
- [Background] FOLDES FF, McNALL PG. 2-Chloroprocaine: a new local anesthetic agent. Anesthesiology. 1952 May;13(3):287-96. doi: 10.1097/00000542-195205000-00009. No abstract available. PMID 14933832
- [Background] Yoos JR, Kopacz DJ. Spinal 2-chloroprocaine: a comparison with small-dose bupivacaine in volunteers. Anesth Analg. 2005 Feb;100(2):566-572. doi: 10.1213/01.ANE.0000143356.17013.A1. PMID 15673895
- [Background] Gonter AF, Kopacz DJ. Spinal 2-chloroprocaine: a comparison with procaine in volunteers. Anesth Analg. 2005 Feb;100(2):573-579. doi: 10.1213/01.ANE.0000143380.36298.4A. PMID 15673896
- [Background] Casati A, Fanelli G, Danelli G, Berti M, Ghisi D, Brivio M, Putzu M, Barbagallo A. Spinal anesthesia with lidocaine or preservative-free 2-chlorprocaine for outpatient knee arthroscopy: a prospective, randomized, double-blind comparison. Anesth Analg. 2007 Apr;104(4):959-64. doi: 10.1213/01.ane.0000258766.73612.d8. PMID 17377114
- [Derived] Guntz E, Jeanne G, Gouwy J, M'rini M, Saxena S, Fils JF, Kapessidou Y. Influence of height on ED95 of intrathecal 2-chloroprocaine for knee arthroscopy: A prospective dose-response clinical trial. Eur J Anaesthesiol. 2022 Jul 1;39(7):602-610. doi: 10.1097/EJA.0000000000001692. Epub 2022 Jun 10. PMID 35695753